CLINICAL TRIAL: NCT06891625
Title: Acute Effects of Spinal Manipulative Therapy, Exercise Therapy and Open-label Placebo on Movement Performance in Individuals With Chronic Back Pain
Brief Title: Movement Performance in Persons With Chronic Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Stiftelsen Rönnbäret (Unknown)
Responsible Party: Principal Investigator, Wilhelmus Grooten, University lecturer, Karolinska Institutet
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2024-07604-01
Record Dates: First submitted 2025-03-06; First posted 2025-03-24 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Chronic Low-back Pain; Back Disorder
Keywords: chiropractic; physical therapy; open-label placebo; motion capture; acute effects; pain-intensity
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: All participants receive all treatments: SMT, MET and OLP
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Spinal manipulation therapy (SMT) (Experimental): Chiropractic treatment
  Interventions: Other: ET; Other: OLP
- Exercise Therapy (ET) (Experimental): Physical therapy treatment
  Interventions: Other: SMT; Other: OLP
- Open Placebo (OLP) (Placebo Comparator): Open-label treatment
  Interventions: Other: SMT; Other: ET

INTERVENTIONS:
Other: SMT — In the present study, a short examination of the whole spine and pelvic area will be performed to identify those segments with the highest restricted range of motion compared to other parts. A standard HVLA manipulation of this area is applied, which refers to Maitland grade 5.
  Arms: Exercise Therapy (ET); Open Placebo (OLP)
Other: ET — In the present study, the participant will, after short warming up, perform three standard exercises aiming to increase the possibility for a person with back pain to control the full range of spinal, pelvis and hip joints (Exercise 1) to increase the motor control and coordination of the muscles controlling the low back, pelvis and hip joints in flexion and rotation (Exercise 2), and to increase the motor control of muscles controlling the low back, pelvis and hip joints in extension (Exercise 3).
  Arms: Open Placebo (OLP); Spinal manipulation therapy (SMT)
Other: OLP — In the present study, the procedure will follow the study of Carvalho, et al. (2016).28 The researcher explains clearly in a positive way to the participants that i) a placebo effect can be powerful, ii) the body can automatically respond to taking placebo pills like Pavlov's dogs that salivated when they heard a clock, iii) that a positive attitude can be helpful, but is not necessary, and iiii) the researcher shows a short video clip (1 minute 25 seconds) of a news report, where participants in an OLP study are interviewed on the positive effects they experienced (https://www.youtube.com/watch?v=Jp14Lhl0T9). Thereafter, the participants are asked to take two pills, containing the inactive substance microcrystalline cellulose from a container clearly labeled with "placebo".
  Arms: Exercise Therapy (ET); Spinal manipulation therapy (SMT)

SUMMARY:
The goal of this laboratory-based cross-over randomized controlled study is to study the immediate effects Spinal manipulative therapy (SMT) and exercise therapy (ET) compared to open-label placebo (OLP) on movement performance, gait, active trunk mobility and pain-intensity in persons with chronic non-specific back pain.

The main question this study aims to answer is: What are the immediate and measurable effects of SMT and ET on work movements, gait, active trunk mobility and pain-intensity in people with chronic non-specific back pain, compared with and in combination with open-label placebo treatment (OP)?

The investigators hypothesize that the participants, after SMT and ET, will perform the lifting task faster, and use more range of motion in most of the joints. They also believe that a greater range of motion is used during gait and that the active ROM in the back is increased, while the pain intensity scores decrease after these interventions. The investigators hypothesize that the control intervention (OLP) could be effective as an add-on intervention, but not as a single intervention.

All participants will receive all three interventions SMT, ET and OLP and to study the immediate effects, the participants will be asked:

* to lift a box with two different weights
* to walk straight forward with and without a cognitive dual task
* perform two clinical tests of active range of motion (
* rate the intensity of their pain "right now"
* rank the treatment effects of these three treatment methods

DETAILED DESCRIPTION:
The occurrence of chronic non-specific back pain (CBP) is costly for Western society and most persons with CBP are functionally limited in their everyday movements. Studies show positive subjective short-term effects after a period of both spinal manipulative therapy (SMT) and exercise therapy (ET), but the immediate effects on of one session SMT/ET on movement performance are unknown. Open placebo is a relatively new field of research and a promising form of treatment for people with nonspecific pain conditions.

The goal of this laboratory-based cross-over randomized controlled study is to study the immediate effects Spinal manipulative therapy (SMT) and exercise therapy (ET) compared to open-label placebo (OLP) on movement performance, gait, active trunk mobility and pain-intensity in persons with chronic non-specific back pain.

Participants with long-term back pain will be recruited through primary care, such as health centers, private clinics and occupational health services.

All participants will receive all three interventions (around 5-8 minutes each)

* SMT: a doctor of chiropractic will perform HVLA spinal manipulation of areas with restricted range of motion.The areas of interest can be from the neck to the pelvis and hips.
* ET: The participants will be asked to perform mobility and motor control exercises of the trunk and pelvic muscles under supervision.
* OLP: The participant takes two pieces of orange gelatin capsules filled with the inactive substance microcrystalline cellulose, following the procedure described in Carvalho et al (2016). In short, participants will be informed that the pills are placebos and will be shown a news report featuring patients with non-specific complaints, such as migraines and irritable bowel syndrome, who describe their positive experiences with placebo.

Movement performance will be studied in an advanced movement analyses laboratory (Qualisys) and operationalized using kinematic parameters such as movement time, relative phase time, range of motion in the spine and adjacent joints, inter-segmental coordination, etc.

To study the immediate effects on movement performance, the participants will be asked to perform the following functional movements before and immediately after each intervention:

* lifting a box with two different weights from just above ground level and place it on a table in front of them
* walking straight forward at a self-selected walking speed with and without a cognitive dual task
* two clinical tests of active range of motion (modified finger-to-floor test, and the modified m-Schober's test)

Moreover, the participants are asked to:

* rate the intensity of their pain "right now" on an 11-point standard numerical rating scale (NRS)

At the end of the experiment, when all interventions have been applied, the participants are asked to:

* rank the treatment effects of these three treatment methods based on their effectiveness, willingness and preference

ELIGIBILITY:
Inclusion Criteria:

* Persons who have either experienced continuous or recurring back pain for a period longer than 3 months). Back pain is defined as problems/discomfort from the spine Th1-S1 with associated costovertebral joints and sacroiliac joints, thus including both the lumbar spine and the thoracic spine. The area of pain extends from Th1 to the inferior gluteal fold but does not include the shoulder blades
* >18 years old,
* those who can speak and understand Scandinavian or English.

Exclusion Criteria:

* "red flags"
* persons with specific back problems, rheumatic inflammatory joint- and/or back diseases, fractures, diagnosed hip osteoarthritis, fibromyalgia, or neurological co-morbidity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Lifting performance | Immediately after each intervention, the participants perform the lifting task. The results will be compared to the baseline measures.
  Participants are asked to perform the movement at a comfortable self-selected speed. They perform two consecutive lifts and between the lifts, the test staff will the object to its original position. To standardize the test, the height of the table is adjusted to 50% of the participant's body height and the horizontal distance between the participant and the table to 75% of his/her arm length. The lift is performed in two situations: one "light" situation and one "moderate/heavy" situation.
  Kinematic and kinetic variables defining movement performance during the lifting task will be used to analyze the data. The lifts will be divided into two phases: a downward and an upward phase, and expressed in % movement-time. For each phase, we will study variables such as fixed time, speed of movement, ROM, intersegmental coordination.

SECONDARY OUTCOMES:
Gait - 1) Temporal gait parameters | Immediately after each intervention, the participants perform the gait task. The results will be compared to the baseline measures.
  The participants are asked to walk straight forward at a self-selected walking speed for about 10 meters. The participants' gait is also studied after the instruction to walk as fast as possible (but not run).
  Gait will be analyzed with temporal gait parameters, such as total cycle time and time in sub-phases. The unit that will be used is milliseconds (ms) and expressed in % of the whole gait cycle, e.g. % single stance, % double support, etc.
Gait - 2) Spatial gait parameters | Immediately after each intervention, the participants perform the gait task. The results will be compared to the baseline measures.
  The participants are asked to walk straight forward at a self-selected walking speed for about 10 meters. The participants' gait is also studied after the instruction to walk as fast as possible (but not run).
  Gait will be analyzed with spatial gait parameters, such as step length and step width, stride length. The SI-unit that will be used is meters (m).
Gait - 3) Joint angles during gait | Immediately after each intervention, the participants perform the gait task. The results will be compared to the baseline measures.
  The participants are asked to walk straight forward at a self-selected walking speed and after an instruction to walk as fast as possible for about 10 meters (but not to run). The subject will be asked to perform these tasks two consecutive times, and the second trial will be used in the analyses.
  Spatial angles (unit: degrees) in neck, upper back, lower back, hips, knees and ankle joints will be analyzed during each gait cycle in three planes: sagittal, frontal and transversal plane. These will be printed vs gait-cycle % and compared to normal values (available from the software). Moreover, angle velocity and inter-segmental coordination, i.e. the movement performance of different segments simultaneously is studied by plotting angle-angle diagrams for an analysis of movement quality.
m-FTF | Immediately after each intervention, the participants perform the test of active range of motion. The results will be compared to the baseline measures.
  Modified finger-to-floor test (m-FTF). Participants will be asked to make an attempt to bend forward as far as possible, keeping their knees, arms, and fingers fully extended. The vertical distance between the tip of the third finger and the floor is measured by placing a ruler under the third finger at a 90° angle to the tape measure on the wall; less distance indicates greater active trunk mobility.
mm-Schober's test | Immediately after each intervention, the participants perform the test of active range of motion. The results will be compared to the baseline measures.
  The modified modified-Schober's test (mm-Schober). Participants will be asked to stand in a neutral position. The examiner will place the thumbs on the subject's spina iliaca posterior superior (SIPS) and a line (lower landmark) is drawn along the midline of the lumbar spine horizontally to the SIPS.While the examiner holds the tape firmly against the subject's skin, he/she marks a second line 15 cm above the first line (upper landmark). Then the subject is asked to make an active forward bend of the trunk without increased pain. The difference between the lines is then measured, and rounded to the nearest mm. The test is positive if the difference between the neutral and flexed position in mm-Schober is less than 5 cm.
Pain-Intensity | Immediately after each intervention, the participants rate their pain-intensity ("pain right now"). The results will be compared to the baseline measures.
  Participants are asked to rate the intensity of their pain "right now" on an 11-point standard numerical rating scale (NRS). They are asked to select one number by filling in a questionnaire, or verbally answering a spoken question such as 'Please tell me which of the numbers from 0 to 10 best describes your pain now'. The scale consists of a horizontal with the words 'no pain' and 'worst possible pain' at either end and lines between the numbers '0' and '10' and includes evenly spaced vertical bars numbered '1' to '9'.
Preference | Immediately after all interventions, the participants evaluate the interventions.
  A final subjective evaluation of the three interventions will be performed by asking the participants to rank the treatment effects of these three treatment methods based on their effectiveness, willingness and preference. Effectiveness will be rated on an 11-point scale (0: not effective/harmful, 10: very effective). Similarly, willingness to use the intervention will be rated starting at " not at all" (0) ranging to "always" (10), and preference will be rated by asking the participants to order the treatments from "best" (1) to "worst" (3). For this three ranking rules are needed: 1) The participants must assign a unique rank to each treatment. 2) There must be one treatment rated as the best (rank 1), one as second best (rank 2), and one as the worst (rank 3). 3) Participants cannot give the same rank to more than one treatment; each treatment has a distinct rank.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Huddinge, Sweden

IPD SHARING:
Plan to Share IPD: Yes
All data will be coded making it impossible to identify individuals. On request, this coded data can be shared.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 10 years after publication
Access Criteria: Researcher or university